CLINICAL TRIAL: NCT05100433
Title: Effect of Passive Ultrasonic Irrigation on Bacteria That Persist After Root Canal Preparation in Teeth With Apical Periodontitis
Brief Title: Effect of Passive Ultrasonic Irrigation on Bacteria That Persist After Root Canal Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ericka Tavares Pinheiro, Associate Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAPESP 2016/15473-0-2
Record Dates: First submitted 2021-09-20; First posted 2021-10-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microbiological analysis of root canals after endodontic procedures (Experimental): Bacterial levels and activity in root canal samples after chemomechanical procedures and ultrasonic irrigation.
  Interventions: Procedure: Ultrasonic irrigation

INTERVENTIONS:
Procedure: Ultrasonic irrigation — Ultrasonic irrigation will be used as a complementary step to chemomechanical procedures to test whether it can improve root canal disinfection.

SUMMARY:
This study aims to evaluate the effectiveness of ultrasonic irrigation in improving root canal disinfection after chemomechanical procedures.

DETAILED DESCRIPTION:
Although chemomechanical procedures promote a drastic bacterial reduction, many root canals remain infected, which points to the need for complementary procedures to improve root canal disinfection. Thus, this clinical study aims to evaluate the effect of passive ultrasonic irrigation as a supplementary disinfection procedure after root canal preparation. Microbiological samples of the root canals of 30 single-rooted teeth with apical periodontitis will be taken at different stages of the endodontic treatment: before preparation (S1), after chemomechanical procedures (S2) and after passive ultrasonic irrigation (S3). The samples will be submitted to the quantitative polymerase chain reaction for bacterial quantification and to the reverse transcription quantitative polymerase chain reaction for bacterial activity analysis. Data will be analyzed using the Wilcoxon test for paired samples (p < 0.05).

ELIGIBILITY:
Inclusion Criteria:

* Teeth with necrotic pulps and asymptomatic apical periodontitis

Exclusion Criteria:

* patients who had received antibiotics during the previous 3 months or had any general disease,
* teeth that could not be properly isolated with rubber dam,
* non-restored teeth,
* periodontal pockets depths greater than 4 mm,
* previous endodontic treatment,
* open apex,
* crown/root fracture
* root resorption or calcifications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Bacterial Activity | through study completion, an average of 3 years
  The metabolic activity of total bacteria in root canal samples after ultrasonic irrigation

SECONDARY OUTCOMES:
Bacterial Levels | through study completion, an average of 3 years
  Quantitative data of total bacteria determined by quantitative polymerase chain reaction after endodontic procedures

CONTACTS AND LOCATIONS:
Locations (1):
- University of São Paulo, São Paulo, São Paulo, Brazil